CLINICAL TRIAL: NCT04475952
Title: Early Diagnosis of Upper Digestive Tract Disease
Acronym: E-DIGEST
Status: Recruiting | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: IRAS 257483
Record Dates: First submitted 2020-07-14; First posted 2020-07-17 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Squamous Cell Carcinoma; Breath Test; Digestive System Disease; Diagnose Disease
MeSH Terms: conditions — Carcinoma, Squamous Cell; Digestive System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oropharyngeal squamous cell carcinoma
- Oesophageal squamous cell carcinoma
- Control

SUMMARY:
Upper digestive tract cancer (UDC) is a major disease burden worldwide encompassing all cancers involving the digestive tract (from oral cavity to duodenum). A majority of patients presenting with this disease are diagnosed late and have poor overall survival rates (<20%). NICE referral guidelines for diagnostic endoscopy are usually associated with late disease. Exhaled breath testing is a non-invasive and acceptable technology utilising mass spectrometry (MS) which has shown promise at diagnosing cancer at an early stage.

Previous research has shown that products formed as a result of metabolism can be measured in breath and saliva (biomarkers). This has the ability to accurately identify patients with upper gastrointestinal (UGI) cancers from breath. Our initial pilot data has demonstrated that changes in the breakdown of metabolites release volatile organic compounds (VOC) which can be measured with MS. This data is supported by other patient studies. However no previous study has been performed utilising a non-invasive technique with breath and saliva. Thus the aim of this study is to identify VOCs present in patients with this disease.

In this multi-centre study the investigators want to overcome the limitations of previous work by utilising non-invasive samples (breath, saliva and urine) in patients in multiple sites. The investigators aim to conduct a study in patients with UDC and those without. The investigators hope that the results of this study will provide evidence for large scale analysis of patients with this disease, demonstrate the feasibility of this technique and move this valuable test forward into mainstream medical practice. The major advantage of this test is that it is easy to undertake and painless for the patient. This study of products in breath, saliva and urine will be useful for detecting UDC to allow treatment at an early stage, improving overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Any patient who:

  * is ≥ 18 years old and below 90 years of age, AND:
  * is undergoing endoscopy as part of their routine clinical care, OR:
  * is undergoing surgical resection of orodigestive tract disease as part of their routine clinical care, OR:
  * is undergoing treatment of orodigestive tract disease as part of their routine clinical care

Exclusion Criteria:

* Any patient who:

  * Lacks capacity or is unable to provide informed consent.
  * Any patient below 18 years of age or over 90 years of age.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients recruited from secondary care will have been referred by their responsible clinician to undergo either a laryngoscopy (which involves visualisation of the highest part of the oesophagus, larynx and vocal cords, upper gastrointestinal endoscopy (which involves a telescope test to visualise the oesophagus, stomach and duodenum) or a lower gastrointestinal endoscopy (which involves a telescope test to visualise the colon) or surgery. No other investigations will be required.
Sampling Method: Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2019-09-13 (Actual); Primary Completion 2025-09-13 (Estimated); Study Completion 2025-09-13 (Estimated)

PRIMARY OUTCOMES:
Non-invasive testing | 5 years
  Samples such as exhaled breath, urine, saliva, tissue and blood will be obtained from patients. These will be analysed with mass spectrometry to identify the compounds changed in patients with the target disease and those without.

CONTACTS AND LOCATIONS:
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No